CLINICAL TRIAL: NCT06319391
Title: Analysis of the Effect of Donor CYP3A5 Gene Polymorphism on Early Tacrolimus Concentration and Postoperative Acute Renal Injury After Liver Transplantation
Status: Active, not recruiting | Type: Observational
Sponsor: Ziqiang Li (Other)
Responsible Party: Sponsor-Investigator, Ziqiang Li, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: JSZ007
Record Dates: First submitted 2024-03-05; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Complete and Accurate Statistical Data of 60 Patients; CYP3A5*3 Genotypes of 60 Donors and Recipients Were Analyzed Accurately; Postoperative Tacrolimus Concentrations Were Accurately Recorded in 60 Patients; According to the Diagnosis and Grading Criteria of Acute Kidney Injury, the Cases and Grading of Postoperative Acute Kidney Injury in 60 Patients Were Counted; Scientific and Rigorous Statistical Analysis of Data
Keywords: CYP3A5; gene polymorphism; tacrolimus; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- donor/acceptor expression group
  Interventions: Other: CYP3A5*1*、CYP3A5*1*3
- donor expression/acceptor non-expression
- donor non-expression/acceptor expression
- donor/acceptor non-expression group
  Interventions: Other: CYP3A5*3*3

INTERVENTIONS:
Other: CYP3A5*1*、CYP3A5*1*3 — 2ml of venous blood was drawn and placed in an EDTA anticoagulant tube. Peripheral blood genomic DNA was extracted according to the instructions of the DNA extraction kit.The reaction system was prepared by polymerase chain reaction (PCR) according to the instructions of PCR amplification system. After 25g/L agarose gel electrophoresis, the bands of amplified products were observed under UV lamp. The PCR products were purified by enzymolysis. The purified product was prepared according to sequencing PCR amplification system. After 1min predenaturation at 96℃, denaturation at 96℃ for 30s, annealing at 56 ℃ for 30s and extension at 72℃ for 1 cycle. A total of 25 cycles were performed for sequencing PCR amplification. The amplified products were purified by ethanol precipitation method.
  Groups: donor/acceptor expression group
Other: CYP3A5*3*3 — 2ml of venous blood was drawn and placed in an EDTA anticoagulant tube. Peripheral blood genomic DNA was extracted according to the instructions of the DNA extraction kit.The reaction system was prepared by polymerase chain reaction (PCR) according to the instructions of PCR amplification system.After 25g/L agarose gel electrophoresis, the bands of amplified products were observed under UV lamp. The PCR products were purified by enzymolysis. The purified product was prepared according to sequencing PCR amplification system. After 1min predenaturation at 96℃, denaturation at 96℃ for 30s, annealing at 56 ℃ for 30s and extension at 72℃ for 1 cycle. A total of 25 cycles were performed for sequencing PCR amplification. The amplified products were purified by ethanol precipitation method.
  Groups: donor/acceptor non-expression group

SUMMARY:
Tacrolimus is the most commonly used immunosuppressant for preventing and treating rejection after liver transplantation. However, its treatment window is narrow, the pharmacokinetic individual differences are large, routine dose according to body weight, sometimes low dose will cause graft rejection of patients, or high dose will lead to infection and liver and kidney toxicity and other adverse reactions. Moreover, the conventional drug testing can not fully reflect the efficacy of tacrolimus, and there are shortcomings of lag, experience and passivity. FK506 is metabolized primarily by cytochrome P450 member 3A5 in the liver and intestines. CYP3A5*3 is the most important factor determining the expression level of CYP3A5. This mutation can cause variable shear and produce unstable protein, so that patients carrying CYP3A5*3/*3 gene do not express CYP3A5. Acute kidney injury is a common and important complication after liver transplantation. Despite recent advances in organ preservation, surgical techniques, and immunosuppressive protocols, the incidence of AKI after orthotopic liver transplantation remains high. AKI has a significant impact on both short - and long-term prognosis of orthotopic liver transplantation recipients. Studies have shown that orthotopic liver transplantation recipients with AKI have significantly higher mortality rates in hospital, at 28 days and at 1 year after surgery than those without AKI. In this study, the relationship between donor and recipient CYP3A5 gene polymorphism and tacrolimus concentration was investigated, and the effect of donor and recipient CYP3A5 gene polymorphism and tacrolimus concentration on acute kidney injury after liver transplantation was investigated. To provide guidance for individual administration of gene-directed tacrolimus in patients, and provide basis for prevention and reduction of postoperative acute kidney injury in liver transplantation patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing orthotopic liver transplantation in our center.
2. The postoperative immunosuppression regimen was tacrolimus、methylprednisolone and balipremumab for injection in all cases,and no drugs that interacted with tacrolimus were used.
3. The postoperative follow-up time was greater than 6 months and no serious rejection occurred during the follow-up period.

Exclusion Criteria:

1. Combined organ transplantation.
2. liver transplant patients on other immunosuppressive regimens.
3. Preoperative CKD or need RRT.
4. Preoperative serum creatinine (SCr) > 133 mol/L.
5. Loss of follow-ups.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 60 patients receiving liver transplantation at the center of Qianfoshan Hospital in 2022.01-2023.06
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Fk506 | 1-28 days postoperatively
  Tacrolimus concentration
Scr | 1-28 days postoperatively
  Reflects indicators of kidney function

CONTACTS AND LOCATIONS:
Overall Officials: Liziqiang Liziqiang, Doctor, Study Director — Party
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital), Jinan, Shandong, China